CLINICAL TRIAL: NCT07154030
Title: Efficacy Of Combined Microneedling Plus Tretinoin 0.025% Or Timolol 0.5% In Treatment Of Stria Rubra
Brief Title: Efficacy Of Combined Microneedling Plus Tretinoin In Treatment Of Stria Rubra
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Kholoud Mostafa Hashem, demonstrator od dermatology, Sohag University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Soh-Med-25-7-7MS
Record Dates: First submitted 2025-08-08; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Striae
Keywords: Timolol; Tretinoin; Stria Rubra; Microneedling
MeSH Terms: conditions — Striae Distensae

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator): microneedling plus tretinoin 0.025%
  Interventions: Procedure: Micro needle injection; Procedure: Micro needle injection only
- Group 2 (Experimental): microneedling plus timolol 0.5%
  Interventions: Procedure: Micro needle injection; Procedure: Micro needle injection only

INTERVENTIONS:
Procedure: Micro needle injection — * Disinfection: the affected area by alcohol 70 %.
  * Topical anaesthetic cream will be applied: pridocaine (lidocaine 2.5% and prilocaine 2.5%) for 30 minutes under occlusion.
  * Microneedling with tretinoin 0.025% of the affected area will be done by dermapen that will be applied on the affected area as follows: inserting the sterilized needle into the dermapen tip, turning on using speed setting and adjusting speed on 5, needle depth of dermapen will be adjusted to (2- 2.5mm) according to the site of the striae, passing vertically over the striae with dermapen in a stamping pattern until pin point bleeding appear.
Procedure: Micro needle injection only — * Disinfection: the affected area by alcohol 70 %.
  * Topical anesthetic cream will be applied: pridocaine (lidocaine 2.5% and prilocaine 2.5%) for 30 minutes under occlusion.
  * Microneedling with timolol 0.5% of the affected area will be done by derma pen that will be applied on the affected area as follows: inserting the sterilized needle into the derma pen tip, turning on using speed setting and adjusting speed on 5, needle depth of derma pen will be adjusted to (2- 2.5mm) according to the site of the striae, passing vertically over the striae with derma pen in a stamping pattern until pin point bleeding appear.

SUMMARY:
Striae distensae (SD), commonly known as stretch marks, are linear dermal scars accompanied by epidermal atrophy . They are often associated with psychological morbidity with a negative impact on quality of life .They are mainly caused by marked stretching in the skin leading to dermal damage and epidermal thinning, leading to linear atrophic scars .

Stretch marks are more common in women , their prevalence in puberty range from 6% to 86% and in obesity, it is 43%. Striae gravidarum (SG), (stretch marks of pregnancy) range between 50% and 90% ,and are more common in younger women.

DETAILED DESCRIPTION:
Striae distensae are most commonly found on the thighs, buttocks, and breasts in girls, and on the lumbosacral area or the outside surface of the thighs in boys. SG appears in the third trimester on the abdomen, breasts or thighs. They are more common in young primigravidae and are linked to higher pregnancy weight, large for gestational age new born, and a higher risk of traumatic vaginal birth .

The SD comes in two forms: striae rubrae (SR) and striae alba (SA). The initial erythematous, stretched flat lesions that are aligned perpendicular to the direction of skin tension represent the acute stage (SR) and they can cause mild itching. The chronic stage (SA) is described when SD have faded and appears atrophic, wrinkled and hypopigmented .

The most common causes of SD include a growth spurt during puberty, pregnancy, positive family history, obesity, and rapid weight gain or loss . Genetic causes including Marfan syndrome, Ehler-Danlos syndrome, and ectodermal dysplasia .

Other causes include cushing disease, anorexia nervosa, infections like T.B and typhoid, chronic liver disease and impaired elastic fibres of dermis. Iatrogenic causes include long term use of topical and systemic steroids and anti-retroviral drugs . Overstretching of the skin lead to dermal damage with inflammatory edema leading to rupture of collagen, elastin and fibronectin. Additionally, there is a defect in fibroblast function, with decrease in fibrillin and elastin production and lack of collagen organization . The treatment modalities for SD range from topical agents to more advanced laser and energy-based devices . Topical treatments such as tretinoin and glycolic acid are widely used for their ability to enhance collagen production and improve skin texture.

Lasers and light devices, particularly fractional CO2 lasers, efficiently promote dermal remodeling and improve the appearance of both SR and SA. No single therapy has emerged as the "gold standard," and combination therapies are recommended . Microneedling as a method of treating stretch marks, stimulates intradermal collagen production , also it can be used as a method of achieving trans-epidermal drug delivery.it also helps elimination of damaged old collagen . Microneedling leads to the release of several growth factors, including platelet-derived growth factors, fibroblast growth factors, and transforming growth factors alpha and beta, which stimulate the migration and proliferation of fibroblasts, producing new collagen and elastin in the papillary dermis. In addition, new capillaries are formed, this neovascularization and neocollagenesis following treatment lead to reduction of scars. The procedure is therefore called "percutaneous collagen induction therapy" .

ELIGIBILITY:
Inclusion Criteria:

* The study will include patients with stria rubra aged ≥18

Exclusion Criteria:

- 1.Pregnant & lactating patients. 2.Patients with bleeding disorders or on anticoagulant therapy. 3.Patients using drugs that exacerbate the striae as systemic corticosteroids in the preceding two months or topical corticosteroid in the preceding one month.

4.Patients having active infection at the treatment area. 5.Patients with keloidal tendency. 6.Patients using other forms of treatment for stria as emollients, glycolic acid peel and laser over the last 2 months.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-09-05 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-09-05 (Estimated)

PRIMARY OUTCOMES:
Evaluate the efficacy of combined microneedling plus tretinoin 0.025% or timolol 0.5% in treatment of stria rubra by noticing gradual changes in the appearance of skin and continuous photographing the site of lesion to notice the physiological changes | 12 months
  Evaluate the efficacy of combined microneedling plus tretinoin 0.025% or timolol 0.5% in treatment of stria rubra by noticing gradual changes in the appearance of skin and continuous photographing the site of lesion to notice the physiological changes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://dx.doi.org/10.4103/ecdt.ecdt_40_23